CLINICAL TRIAL: NCT05103293
Title: Neoadjuvant Therapy for Breast Cancer Based on Patient-derived Tumor-like Cell Clusters Advanced Drug Sensitization Regimens: a Phase II Randomized Controlled Clinical Study
Brief Title: PTC Guiding Neoadjuvant Treatment in Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, YU Xingfei, Doctor, Zhejiang Cancer Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PTC-breastNAT
Record Dates: First submitted 2021-10-06; First posted 2021-11-02 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Pathological Conditions, Signs and Symptoms
Keywords: patient-derived tumor-like cell clusters; breast cancer; neoadjuvant therapy; pathologic complete response
MeSH Terms: conditions — Pathological Conditions, Signs and Symptoms; Breast Neoplasms; Pathologic Complete Response

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTC group (Experimental): Patients randomized into this group receiving PTC test and choose regimens according to this test results
  Interventions: Diagnostic Test: patient-derived tumor-like cell clusters drug sensitivity test
- Control group (No Intervention): Patients randomized into this group receiving routine regimens according to subtypes

INTERVENTIONS:
Diagnostic Test: patient-derived tumor-like cell clusters drug sensitivity test — Intervention Description：Neoadjuvant therapy regimen of patients in the PTC group is guided by PTC drug sensitivity results. After operation, adjuvant targeted therapy for pCR patients is based on original treatment, adjuvant targeted therapy for non-pCR patients is based on a secondary PTC drug sensitivity results.
  Other Names: PTC
  Arms: PTC group

SUMMARY:
Patients with breast cancer meet criteria for enrollment are randomized into PTC group or control group. The neoadjuvant therapy regimens are guided by PTC test in the PTC group. The regimens in control group are included of (dd)EC-T for HER2 negative subtype, TCH(P) or EC-TH(P) for HER2 positive subtype. We compared the pCR rate between two groups as the primary endpoint.

DETAILED DESCRIPTION:
1. Before neoadjuvant therapy, all samples will be obtained by core needle biopsy for PTC drug sensitivity test.
2. After obtaining drug sensitivity results and confirming ER/PR and HER2 expression state, all recruited patients will be randomized into the PTC group or the routine treatment group, according to the method of random number table.
3. Beijing Cornerstone Life Science and Technology Co., Ltd. is responsible for gene sequencing and PTC drug sensitivity test for biological samples. All samples for the study are clinical residuals and will be used in the study, store or destruction is unapplicable.
4. Neoadjuvant therapy regimen in the PTC group is guided by PTC drug sensitivity results, and regimen in the routine treatment group is based on clinical guideline, such as (dd)EC-T for HER2 negative breast cancer, and TCH(P) or EC-TH(P) for HER2 positive breast cancer. All neoadjuvant therapy will be completed before operation if without PD.
5. According to postoperative pathological remission, pCR patients in two groups continued to complete adjuvant targeted therapy based on original treatment. For non-pCR patients in the PTC group, PTC drug sensitivity test will be done again to guide adjuvant therapy, for non-pCR patients in the routine treatment group, Capecitabine for HER2 negative breast cancer, and T-DM1 or H(P) will be selected.
6. All patients will be received radiotherapy or endocrine therapy if necessary.

ELIGIBILITY:
Inclusion Criteria:

1. Female between 18 to 70 years old.
2. Patients diagnosed with invasive breast cancer by pathology.
3. Clinical stage considered as T2-4N0-2M0 .
4. HER2 overexpression by IHC or FISH positive.
5. Patients plan to accept neoadjuvant therapy or plan to accept adjuvant therapy after neoadjuvant therapy and surgery.

Exclusion Criteria:

1. Patients have already accepted any other anti-tumor treatment not included in our project.
2. Patients with metastasis are not considered surgery therapy.
3. Patients cannot accept chemotherapy or anti-HER2 targeted therapy, because of severe cardiovascular diseases or other reasons

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
pCR rate | one month after operation
  pathological complete response
objective response rate | half year after randomize
  cCR or PR or SD according to RECIST1.1

SECONDARY OUTCOMES:
2y-Disease free survival rate | 2year
  survive with neither invasive recurrence nor new invasive diseases
5y-Disease free survival rate | 5year
  survive with neither invasive recurrence nor new invasive diseases

CONTACTS AND LOCATIONS:
Overall Officials: Xingfei Yu, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China